CLINICAL TRIAL: NCT05797077
Title: Postoperation Maintenance Therapy for Resectable Liver Metastases of Colorectal Cancer Guided by ctDNA: a Multicenter, Randomized, Controlled, Phase III Clinical Trial.
Brief Title: Postoperation Maintenance Therapy for Resectable Liver Metastases of Colorectal Cancer Guided by ctDNA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010(PY)2022-10
Record Dates: First submitted 2023-03-20; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Liver Metastases; Circulating Tumor Cell; Cancer, Therapy-Related
Keywords: Colorectal Cancer; Liver Metastases; ctDNA; maintenance therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplastic Cells, Circulating; Neoplasms, Second Primary | interventions — Folfox protocol; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant chemotherapy combined with maintenance therapy (Experimental)
  Interventions: Procedure: Colorectal resection surgery.; Drug: FOLFOX chemotherapy regimen; Drug: Capecitabine
- Single adjuvant chemotherapy (Sham Comparator)
  Interventions: Procedure: Colorectal resection surgery.; Drug: FOLFOX chemotherapy regimen

INTERVENTIONS:
Procedure: Colorectal resection surgery. — Colorectal cancer radical resection combined with liver metastasis resection or ablation.
Drug: FOLFOX chemotherapy regimen — Chemotherapy regimens recommended include oxaliplatin-based CapeOx or FOLFOX regimens, or single-agent 5-FU/LV, capecitabine, or combination with targeted therapy.
  Other Names: CapeOx chemotherapy regimen
Drug: Capecitabine — Maintenance therapy is recommended to be continued with low-toxicity drugs such as 5-FU/LV or capecitabine, and may be combined with targeted therapy. Treatment should be discontinued once ctDNA testing is negative.
  Other Names: 5-FU/LV
  Arms: Adjuvant chemotherapy combined with maintenance therapy

SUMMARY:
The goal of this clinical trial is to compare in resectable liver metastases colorectal cancer patients.The main question it aims to answer is to investigate whether the progression-free survival (PFS) of resectable colorectal liver metastasis (CRLM) patients with positive ctDNA after surgery is superior with the combination of adjuvant chemotherapy and maintenance therapy compared to adjuvant chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females, aged 18-75 years;
2. Patients with liver metastatic colorectal cancer who have undergone R0 resection based on MDT evaluation (including patients whose metastases have been treated with ablation achieving similar R0 resection effect);
3. Postoperative ctDNA-positive patients;
4. ASA grade < IV and/or ECOG performance status score ≤ 2;
5. Participants must have a full understanding of the study and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Patients with distant metastases to other sites, including the pelvis, ovaries, peritoneum, etc.
2. Patients with a history of other malignant tumors.
3. Patients with severe liver or kidney dysfunction, cardiorespiratory dysfunction, coagulation dysfunction, or underlying diseases that cannot tolerate chemotherapy.
4. Patients who are allergic to any component of the study.
5. Patients who have received other tumor-related investigational drug treatments.
6. Patients with severe uncontrolled recurrent infections or other severe uncontrolled accompanying diseases.
7. Patients with other factors that may affect the study results or lead to early termination of the study, such as alcoholism, drug abuse, other serious diseases requiring comprehensive treatment (including mental illness), and severe laboratory abnormalities.
8. Patients with a history of severe mental illness.
9. Pregnant or lactating women.
10. Patients who, in the opinion of the researchers, have other clinical or laboratory conditions that make them unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2029-02-20 (Estimated); Study Completion 2031-02-20 (Estimated)

PRIMARY OUTCOMES:
3-years Progression Free Survival | 3 years after operation.
  PFS is defined as the time from randomization to the occurrence of any progression or death from any cause.
5-years Progression Free Survival | 5 years after operation.
  PFS is defined as the time from randomization to the occurrence of any progression or death from any cause.

SECONDARY OUTCOMES:
3-years overall survival | 3 years after operation.
  Overall survival is defined as the time from randomization to death from any cause. For patients who are still alive at the time of the final analysis, the date of the last contact will be recorded.
5-years overall survival | 5 years after operation.
  Overall survival is defined as the time from randomization to death from any cause. For patients who are still alive at the time of the final analysis, the date of the last contact will be recorded.
Complication | 5 years.
  he complications of adjuvant therapy usually refer to the adverse events that occur during or after treatment, including but not limited to chemotherapy-related adverse reactions, radiation therapy-related adverse reactions, and postoperative complications. Specifically, chemotherapy-related adverse reactions may include nausea, vomiting, diarrhea, anemia, and infections; radiation therapy-related adverse reactions may include skin inflammation, nausea, vomiting, diarrhea, fatigue, and dry mouth; postoperative complications may include bleeding, infection, intestinal obstruction, and poor wound healing. Researchers typically record the types, severity, and impact of these complications on treatment to evaluate the safety and tolerability of adjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided